CLINICAL TRIAL: NCT07116239
Title: Steady-state Pharmacokinetics and Pharmacodynamics of Edoxaban in Adults With Nephrotic Syndrome: A Non-randomized Open-label, Parallel Arm and Single-center Study
Brief Title: Edoxaban Steady-State PK/PD in Adults With Nephrotic Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Collaborators: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2025-h009
Record Dates: First submitted 2025-07-25; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Nephrotic Syndrome; Hypoalbuminemia
Keywords: edoxaban; nephrotic syndrome; hypoalbuminemia; enoxaparin
MeSH Terms: conditions — Nephrotic Syndrome; Hypoalbuminemia | interventions — edoxaban; Enoxaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Edoxaban NS Group 1 (Experimental): Patients with mild hypoalbuminemia (serum albumin >25g/L and <30g/L), taking edoxaban 60mg orally once daily
  Interventions: Drug: Edoxaban 60 mg
- Edoxaban NS Group 2 (Experimental): Patients with severe hypoalbuminemia (serum albumin ≤25g/L), taking edoxaban 60mg orally once daily
  Interventions: Drug: Edoxaban 60 mg
- LMWH NS Group 1 (Active Comparator): Patients with mild hypoalbuminemia (serum albumin >25g/L and <30g/L), injecting enoxaparin sodium 0.4ml subcutaneously once daily
  Interventions: Drug: Enoxaparin 40 mg
- LMWH NS Group 2 (Active Comparator): Patients with severe hypoalbuminemia (serum albumin ≤25g/L), injecting enoxaparin sodium 0.4ml subcutaneously once daily
  Interventions: Drug: Enoxaparin 40 mg
- Healthy Volunteer Group (Other): Healthy volunteers, taking edoxaban 60mg orally once daily
  Interventions: Drug: Edoxaban 60 mg

INTERVENTIONS:
Drug: Edoxaban 60 mg — film-coated tablet, manufactured by Daiichi Sankyo Europe GmbH
  Other Names: LIXIANAN
  Arms: Edoxaban NS Group 1; Edoxaban NS Group 2; Healthy Volunteer Group
Drug: Enoxaparin 40 mg — enoxaparin sodium, prefilled syringe of 0.4mL injectable solution, manufactured by SANOFI WINTHROP INDUSTRIE
  Other Names: CLEXANE
  Arms: LMWH NS Group 1; LMWH NS Group 2

SUMMARY:
A study to evaluate the impact of nephrotic syndrome on the steady state pharmacokinetics and pharmacodynamics of edoxaban compared to health volunteers, and whether edoxaban can provide an equivalent anticoagulant effect to enoxaparin sodium.

ELIGIBILITY:
Inclusion Criteria:

1. Nephrotic syndrome Group:

   * Age between 18-70 years old
   * Diagnosed with nephrotic syndrome: proteinuria≥3.5 g/24h or morning urine protein/creatinine ratio ≥3.0g/g), with serum albumin <30g/L present at the time of enrollment, with or without edema or hyperlipidemia
   * Calculated creatinine clearance (CrCl) >50ml/min using the Cockcroft-Gault formula
   * Actual body weight >60kg, and body mass index within the range of 18.5-28kg/m2
   * Signed informed consent form
2. Healthy volunteer Group:

   * Age between 18-70 years old
   * Serum albumin ≥40g/L
   * Calculated CrCl >50ml/min using the Cockcroft-Gault formula
   * Actual body weight >60kg, and body mass index within the range of 18.5-28kg/m2
   * Signed informed consent form

Exclusion Criteria:

* Serun albumin <30 g/L for other reasons in patients with nephrotic syndrome as judged by the investigator
* Prolonged PT, INR, APTT at baseline (defined as greater than the upper limit of normal values)
* Platelet count <100×109/L or ≥300×109/L due to hematological diseases confirmed by laboratory tests
* History of: gastrointestinal bleeding, intracranial hemorrhage, hemoptysis, or other clinically documented bleeding from internal organs within the last 3 months; surgery (except >3 days after renal biopsy without bleeding complications) or trauma. Bleeding complications after renal biopsy are defined as: ① bleeding (hematuria, perirenal hematoma, or arteriovenous fistula) that occur after renal biopsy requiring transfusion, resulting in altered hemodynamics, or requiring surgery or interventional treatment; ② symptomatic perirenal hematoma; and ③visible hematuria that persist for >3 days postoperatively.
* A lesion or condition with a significant risk of major bleeding, such as current or recent gastrointestinal ulcer, malignant tumors with a high risk of bleeding, esophageal varices, arteriovenous malformations, vascular aneurysms, or major intravertebral or intracerebral vascular malformations.
* Serious bleeding disorders as judged by the investigator
* Systemic lupus erythematosus with or without renal damage
* Bleeding or thrombophilia disorders as judged by the investigator
* History of stroke
* History of congestive heart failure (New York grade II or above) at the time of screening
* Liver dysfunction (cirrhosis or bilirubin >2×, and serum transaminases >3×, upper limit of normal)
* Use of (but not limited to) the prescription medications that are inhibitors or inducers of CYP3A4 and/or P-gp within the past 14 days:

  * CYP3A4 inducers (e.g., rifampicin, carbamazepine, phenytoin, etc.) ②CYP3A4 inhibitors (e.g., ketoconazole, ritonavir, clarithromycin, etc.)

    * P-gp inducers (e.g., apalutamide, rifampicin, etc.) ④ P-gp inhibitors (e.g., dronedarone, cyclosporine, erythromycin, ketoconazole, quinidine, verapamil, amiodarone, etc.) ⑤Selective serotonin reuptake inhibitors (SSRI) or serotonin-norepinephrine reuptake inhibitors (SNRI)
* Use of antiplatelet and/ or anticoagulant agents within 5 half-lives (at least 7 days): including but not limited to heparin, heparin derivatives, aspirin, clopidogrel, prasugrel, nonsteroidal anti-inflammatory drugs, warfarin, rivaroxaban, dabigatran, apixaban, etc.
* Pregnant or breastfeeding women or women of childbearing age without contraception
* Uncontrolled severe hypertension (SBP≥180mmHg, DBP≥110mmHg)
* Conditions considered unsuitable for inclusion in this study, judged by investigator
* Patients with hypersensitivity to the active ingredient or other excipients of the Edoxaban and enoxaparin sodium
* History of immune-mediated heparin-induced thrombocytopenia (HIT) or presence of circulating antibodies within the previous 100 days.
* Spinal or epidural anesthesia or local anesthesia within 24 hours prior to the administration of enoxaparin sodium and Edoxaban

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
area under the steady-state plasma concentration-time curve (AUCss) | Day 4 post-administation
  ① Steady-state PK parameters of edoxaban in nephrotic syndrome patients versus healthy volunteers: area under the steady-state plasma concentration-time curve (AUCss)
time to peak (Tmax) | Day 4 post-administation
  Steady-state PK parameters of edoxaban in nephrotic syndrome patients versus healthy volunteers: time to peak (Tmax)
trough concentration at steady state (Css_min) | Day 4 post-administation
  Steady-state PK parameters of edoxaban in nephrotic syndrome patients versus healthy volunteers: trough concentration at steady state (Css_min)
peak concentration at steady state (Css_max) | Day 4 post-administation
  Steady-state PK parameters of edoxaban in nephrotic syndrome patients versus healthy volunteers: peak concentration at steady state (Css_max)
elimination half-life (t1/2) | Day 4 post-administation
  Steady-state PK parameters of edoxaban in nephrotic syndrome patients versus healthy volunteers: elimination half-life (t1/2)
average steady-state plasma concentration (Css_av) | Day 4 post-administation]
  Steady-state PK parameters of edoxaban in nephrotic syndrome patients versus healthy volunteers: average steady-state plasma concentration (Css_av)
apparent volume of distribution (Vd/F) | Day 4 post-administation
  Steady-state PK parameters of edoxaban in nephrotic syndrome patients versus healthy volunteers: apparent volume of distribution (Vd/F)
clearance (CL/F) | Day 4 post-administation
  Steady-state PK parameters of edoxaban in nephrotic syndrome patients versus healthy volunteers: clearance (CL/F)
anti-FXa activity | Day 4 post-administation
  Steady-state PD parameters of edoxaban versus enoxaparin in nephrotic syndrome patients: anti-FXa activity
prothrombin time (PT) | Day 4 post-administation
  Steady-state PD parameters of edoxaban versus enoxaparin in nephrotic syndrome patients: prothrombin time (PT)
activated partial thromboplastin time(APTT) | Day 4 post-administation
  Steady-state PD parameters of edoxaban versus enoxaparin in nephrotic syndrome patients: activated partial thromboplastin time(APTT)
antithrombin Ⅲ(AT-III) | Day 4 post-administation
  Steady-state PD parameters of edoxaban versus enoxaparin in nephrotic syndrome patients: antithrombin Ⅲ(AT-III)
Protein C | Day 4 post-administation
  Steady-state PD parameters of edoxaban versus enoxaparin in nephrotic syndrome patients: Protein C
Protein S | Day 4 post-administation
  Steady-state PD parameters of edoxaban versus enoxaparin in nephrotic syndrome patients: Protein S
D-Dimer | Day 4 post-administation
  Steady-state PD parameters of edoxaban versus enoxaparin in nephrotic syndrome patients: D-Dimer

OTHER OUTCOMES:
Safety Assessment | from the date of informed consent form signature to day 8 post-administration
  Adverse events will be collected and coded according to the Medical Dictionary for Regulatory Activities (MedDRA)